CLINICAL TRIAL: NCT01820221
Title: Staples Compared With Subcuticular Suture for Skin Closure After Cesarean Delivery in Obese Patients
Brief Title: Sutures vs. Staples Skin Closure After C-section in Obese Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment and Pi had no time.
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 138350
Record Dates: First submitted 2013-03-19; First posted 2013-03-28 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Obesity; Pregnancy
Keywords: cesarean delivery; wound complications; skin closure methods
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: Skin closure with suture (Active Comparator): Subjects in this group will be randomized to suture for skin closure with computer generated random card draw.
  Interventions: Procedure: Suture vs. staples closure method after c-section in obese women.
- Arm 2: Skin closure with staples (Active Comparator): Subjects randomized to skin closure with staples with computer generated random card draw.
  Interventions: Procedure: Suture vs. staples closure method after c-section in obese women.

INTERVENTIONS:
Procedure: Suture vs. staples closure method after c-section in obese women. — Random card draw to either suture skin closure or staple skin closure arm of study.

SUMMARY:
This is a randomized prospective clinical trial designed to determine the wound complication rates for stainless steel staples versus subcuticular suture for skin closure in the obese parturient (BMI≥ 30kg/m2) undergoing cesarean delivery.

ELIGIBILITY:
Inclusion criteria:

* 18 years or older
* BMI ≥ 30kg/m2 on admission to labor and delivery
* Patient is for scheduled cesarean delivery or in non-emergent labor but has an indication for cesarean delivery
* Singleton pregnancies
* Gestational age ≥ 24weeks
* Cesarean delivery performed under regional anesthesia

Exclusion criteria:

* Refusal to participate
* BMI < 30kg/m2
* < 24 weeks gestation
* Intrauterine fetal demise
* Chronic pain syndrome requiring chronic narcotic use
* Emergent clinical situations which preclude obtaining informed consent

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 148 (Actual)
Dates: Start 2013-03; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Wound complication rates | 6 weeks postpartum
  Wound complications will be classified as minor and major and the major complications will be further stratified as Seroma, Hematoma and Wound Infection/Surgical site infection (SSI).
  1. Minor wound disruption: any wound disruption that DOES not require that the incision be opened, evacuated, irrigated or debrided. There is no evidence of infection including erythema, induration or purulent material. No antibiotic therapy is given.
  2. Major wound disruption requires that incision be opened, evacuated, and or irrigated or debrided and includes:
     * Seroma: collection of serous fluid in the wound without evidence of infection
     * Hematoma: Demonstrable blood clot between the rectus fascia and the skin
     * Infection: Any wound that drains purulent material and shows at least 2 of the classic signs of infection; induration, erythema, tenderness, fever. Wound infections will be further classified as superficial or deep.

SECONDARY OUTCOMES:
Post-operative pain | 72 hours postpartum
  To allow for adequate monitoring and assessment of postoperative pain, standardized postoperative pain analgesia protocol at our institution will be followed. This comprises of non-steroidal anti- inflammatory drugs and Narcotics as needed. Patients will be asked to complete a visual analog pain scale ranging from 0-10 on postoperative day 2. Information on use of pain medication during hospitalization and frequency will also be collected from the medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Mary L Racher, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States